CLINICAL TRIAL: NCT07105501
Title: Hidden Auricular Amyloid Deposits and Aortic Stenosis: Clinical and Prognostic Implications in Aortic Valve Replacement Surgery
Brief Title: Atrial Amyloid May Influence Outcomes in Patients Undergoing Surgical Aortic Valve Replacement
Acronym: AORTICMARKER
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CEI: PI-19-031.
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Aortic Stenosis; Amyloid
Keywords: Aortic valve replacement surgery; Amyloid; Atrial deposits; Biomarkers; spatial transcriptomics
MeSH Terms: conditions — Aortic Valve Stenosis; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — A histological biobank with atrial and interventricular septum samples is available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CONGO +: Patients with amyloid deposits in atrial histological samples. As this is an observational study, no intervention was performed on the subcohort, which was defined as CONGO+ based on the presence of amyloid deposits observed in atrial samples collected during surgery.
- CONGO -: Patients without amyloid deposits in atrial histological samples. As this is an observational study, no intervention was performed on the subcohort, which was defined as CONGO- based on the no presence of amyloid deposits observed in atrial samples collected during surgery.

SUMMARY:
Background (Context):

Some older adults who undergo surgery to replace a narrowed heart valve (called aortic stenosis) may also have small protein deposits in their heart. These protein clumps, known as amyloid, are more often found in people with a certain condition called amyloidosis. However, in many cases, these deposits are found only in the upper chambers of the heart (called atria) and without any previous diagnosis of the disease. The meaning and health impact of these hidden amyloid deposits are still unclear.

Objectives (What the investigators wanted to find out):

This study aimed to understand how common these protein deposits are in people with aortic valve disease, what this deposits are made of, and how they affect recovery and health after heart surgery. To do this, various types of analysis were combined, including tissue samples, blood tests, and advanced genetic studies.

Methods (What the investigators did):

Seventy patients undergoing surgery to replace the aortic valve were studied. During the operation, small samples were collected from the top part of the heart and analyzed in the lab using special dyes and microscopes. Substances in blood were also measured, and health status was monitored over the following year. For some samples, advanced genetic tools were used to investigate processes at the level of individual cells.

DETAILED DESCRIPTION:
The study aims to find out whether deposits of amyloid (an abnormal protein that builds up in tissues) in the upper chambers of the heart are linked to worse recovery after aortic valve replacement surgery. For example, it looks at whether these deposits are related to hospital readmissions, irregular heart rhythms, or problems with kidney function after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Signed specific informed consent (see attached).
* Severe aortic stenosis with surgical indication.
* Elective isolated aortic valve replacement surgery via full or partial median sternotomy.

Exclusion Criteria:

* Urgent or emergency surgery (patients in cardiogenic shock, under intra-aortic balloon pump therapy or any other mechanical support, or receiving vasoactive drugs).
* Combined surgery with any additional procedure.
* Ischemic heart disease with significant lesions confirmed by preoperative invasive catheterization, with or without concomitant revascularization during aortic valve replacement surgery.
* Concomitant endocarditis.
* Inability to collect surgical tissue samples. Initially, all patients with at least one histological sample were included; later, only those with both atrial and septal samples were analyzed.
* Extracardiac disease with a life expectancy of less than 365 days.
* Patient with a previous and/or current diagnosis of any form of amyloidosis.
* Surgical access other than full or partial median sternotomy.
* Patients with severe aortic stenosis but with a TAVI indication as decided by a multidisciplinary heart team (including interventional cardiology, clinical cardiology, and cardiac surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study cohort includes consecutive patients who underwent isolated aortic valve replacement at Germans Trias i Pujol Hospital, and who met the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
NT-proBNP levels | From enrollment to the one-year follow-up
  NT-proBNP preoperative and follow-up levels in each group
Metrnl levels | from enrollment to the one-year follow-up
  Metrnl preoperative and follow up levels
New-onset postoperative atrial fibrillation | From enrollment to the one-year follow-up
  New presence of postoperative atrial fibrillation
Hospital readmission | From enrollment to the one - year follow-up
  Hospital readmission in the first year follow-up
Postoperative quality of life | From enrollment to the one-year follow-up
  Use of the EuroQuol subjectives health test preoperatively and at one-year follow-up. The test completed title is EuroQuol 5D-5L (or EQ-5D-5L), and it consists of a final score ranging from 0 to 100 points, with 0 representing the worst possible health and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Ignasi Julià, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- hospital universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT07105501/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT07105501/ICF_001.pdf